CLINICAL TRIAL: NCT00581386
Title: A Randomized Clinical Comparison Of The King Systems Disposable Laryngeal Tube Suction (LTS-D), The Esophageal Tracheal Combitube (ETC) And The Proseal Laryngeal Mask Airway (PLMA) In Adult Patients
Brief Title: Clinical Comparison of the Airway Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Carin A. Hagberg, Professor and Chairman, Joseph C. Gable, MD Endowed Chair, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-04-254
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2010-03-04 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Endotracheal Intubation; Supraglottic Airway
Keywords: Endotracheal Intubation; Supraglottic Airway
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- LTS-D (Experimental): All the cases were divided into one of the group LTS-D, PLMA, and ETC
  Interventions: Device: LTS-D
- ProSeal Laryngeal Mask Airway (Experimental): All patients were divided into either LTS-D, PLMA, or the ETC group.
  Interventions: Device: ProSeal Laryngeal Mask Airway
- Esophageal Tracheal Combitube (ETC) (Experimental): All patients are divided into one of the group, LTS-D, PLMA, or the ETC.
  Interventions: Device: Esophageal Tracheal Combitube (ETC)

INTERVENTIONS:
Device: LTS-D — supra-glottic airway device
  Other Names: LTS-D King Systems, Noblesville, IN
  Arms: LTS-D
Device: ProSeal Laryngeal Mask Airway — pre-existing double-lumen supra-glottic device
  Other Names: Laryngeal Mask Airway (PLMA, LMA North America Inc.)
  Arms: ProSeal Laryngeal Mask Airway
Device: Esophageal Tracheal Combitube (ETC) — disposable double-lumen tube
  Other Names: ETC
  Arms: Esophageal Tracheal Combitube (ETC)

SUMMARY:
The purpose of this study is to evaluate a new supra-glottic airway device, the "Disposable Laryngeal Tube Suction" (LTS-D; King Systems, Noblesville, IN). We propose to test its ease of insertion, position within the airway, patency of drain tube and anatomic sealing properties during spontaneous ventilation in anesthetized patients. The study device will be compared to the ProSeal Laryngeal Mask Airway (PLMA, LMA North America Inc.) and the Esophageal Tracheal Combitube (ETC; Tyco Healthcare/Mallinckrodt Nellcor, Pleasanton, Calif).

DETAILED DESCRIPTION:
During the past decade, several pharyngeal airways have been introduced into clinical practice for airway management, such as the Laryngeal Mask Airway (LMA), the Cuffed Oropharyngeal Airway (COPA), the Esophageal Tracheal Combitube (ETC), and most recently, the Laryngeal Tube (LT). These airway devices have become very popular because of their ability to maintain an airway without perturbing the trachea, and can be used in patients without muscle relaxation and who are only lightly anesthetized.

The LMA generally provides an adequate airway, but certain problems remain. (1) In 8-33% of LMA placements, more than one attempt is required. (2) It is sometimes difficult to advance the LMA without extending the neck (which is contraindicated in some patients). (3) The device does not protect the airway from aspiration of gastric contents. (4) It does not provide an airtight seal around the larynx (the usual pressures causing leakage of gas being 15-20 cm H20). Consequently, the device functions poorly during positive-pressure ventilation. (5) The esophagus is included within the rim of the LMA in 10-15% of patients, directly exposing the esophagus to positive airway pressures. This often results in insufflation of the stomach and postoperative discomfort.

The ETC is a disposable double-lumen tube that combines the features of a conventional endotracheal tube with those of an esophageal obturator airway. It is appropriate for prehospital, intraoperative, and emergency use and is especially useful for patients in whom direct visualization of the vocal cords is not possible, patients with massive airway bleeding or regurgitation, limited access to the airway, and patients in whom neck movement is contraindicated. Ventilation with the ETC is possible with either tracheal or esophageal intubation, as its distal cuff seals off the esophagus to prevent aspiration of gastric contents. The ETC has a 6.9% incidence of placement failure and a failed ventilation rate of 21.1%.

The Laryngeal Tube Suction (LTS; VBM Medizintechnik; King Systems, Noblesville, IN) is a supra-glottic airway device designed to provide a more effective seal than the LMA, thus eliminating problems 3-5 described above. The insertion of the standard laryngeal tube is generally easy. The reported success rate of insertion of, and ventilation through, the laryngeal tube ranges from 92-100% for the earlier prototype and 97-100% for the newest version. It is a flexible, curved tube that passes through the mouth, advances posterior to the epiglottis, and terminates in the upper esophagus. The multi-use, double-lumen, silicon LTS is designed with ventilation outlets located between an oropharyngeal and an esophageal, low-pressure cuff. The second lumen allows for an orogastric tube to be passed through for gastric drainage and pressure release. Patients at risk of regurgitation now have an alternative to tracheal intubation. This device has been used in a number of patients by anesthesiologists in Europe. There are many published scientific abstracts in the use of the LTS. A disposable version of the LTS is now available, the LTS-D. The LTS-D offers the same benefits as the LTS, but being disposable, it also eliminates the risk of cross-infection.

The ProSeal Laryngeal Mask Airway (PLMA, LMA North America Inc.) is the pre-existing double-lumen supra-glottic device that allows gastric drainage and pressure release. Its design is based on the LMA with an added lumen. It is reusable. The ProSeal exhibits an unsuccessful ventilation rate of 9%, and a first time insertion failure of 12.7%. Currently, the ProSeal exhibits a 3% incidence of foldover during insertion that prevents it from functioning properly. Due to differences in design, we postulate that the LTS-D will have a lower incidence of foldover than the PLMA.

This clinical study has been designed to compare the ProSeal, ETC and LTS-D as to the ease of placement and ventilation during controlled ventilation, proper positioning, the seal pressure with each placement, the patency of the drain tube by suctioning and measuring stomach contents, and finally, any complications with their use. Fiberoptic observations through each device will provide information in relation to the epiglottis and the distal opening of the device.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects will be adult surgical candidates aged 18-80, ASA I-III, Mallampati I or II, presenting for elective surgery who require general anesthesia in whom tracheal intubation is not necessary.
2. Both male and female patients will be included.

Exclusion Criteria:

* Patients will be excluded from the study if they present as Mallampati III or IV, ASA IV-V or emergency status. Additionally, they will be excluded if they meet one of the contraindication criteria of the LMA ProSeal including:

  1. Obesity
  2. Pregnancy
  3. History of gastric regurgitation, heart burn, ileus or "full stomach"
  4. History of low pulmonary compliance or high pulmonary resistance
  5. Known history of difficult endotracheal intubation or signs suggesting the possibility of difficult intubation
  6. Pharyngeal pathology or
  7. Upper airway obstruction due to laryngeal pathology.
* Additionally, they will be excluded if they meet one of the contraindication criteria for the Combitube including:

  1. Intact gag reflexes
  2. Height <4 feet
  3. Central airway obstruction
  4. Recent ingestion of caustic substances
  5. Known esophageal pathology, or
  6. Known latex allergy.
* They will also be excluded if any tracheal disease is present such as tracheal tumors, stenosis or previous tracheal surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin A. Hagberg, M.D., Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Memorial Hermann Hospital between 05/30/2007 and 04/15/2009. The patients enrolled were undergoing general anesthesia.
Pre-assignment Details: There were no enrolled participants excluded from trial before assignment to groups.
Groups:
- Disposable Laryngeal Tube Suction (LTS-D): Patients were randomly distributed into this group. The patients assigned to this group were intubated using a new LMA device the LTS-D.
- Esophageal Tracheal Combitube(ETC): Patients were randomly assigned into this group. The patients assisgned to this group were intubated with the device ETC.
- ProSeal Laryngeal Mask Airway (PLMA): Patients were randomly assigned into this group. The patients in this group were intubated with the device PLMA.
Period: Overall Study
Arm/Group | Disposable Laryngeal Tube Suction (LTS-D) | Esophageal Tracheal Combitube(ETC) | ProSeal Laryngeal Mask Airway (PLMA)
Started | 73 (05/30/2007) | 73 (05/30/2007) | 72 (05/30/2007)
Completed | 73 (04/15/2009) | 73 (04/15/2009) | 72 (04/15/2009)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disposable Laryngeal Tube Suction (LTS-D) | Esophageal Tracheal Combitube(ETC) | ProSeal Laryngeal Mask Airway (PLMA) | Total
Number analyzed (Participants) | 73 | 73 | 72 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 73 | 73 | 72 | 218
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.84 (14.95) | 39.45 (13.73) | 40.08 (13.68) | 40.47 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 17 | 63
  Male | 50 | 50 | 55 | 155
Region of Enrollment [Number; unit: participants]
  United States | 73 | 73 | 72 | 218

OUTCOME MEASURES:

1. Primary Outcome: Duration of Intubation
Description: The time taken to successfully place the device in seconds.
Time Frame: duration of intubation
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Disposable Laryngeal Tube Suction (LTS-D) | Esophageal Tracheal Combitube(ETC) | ProSeal Laryngeal Mask Airway (PLMA)
Number analyzed (Participants) | 73 | 73 | 72
seconds | 30.9 (18.7) | 30.8 (23.3) | 30.17 (31.53)

2. Primary Outcome: Number of Participants With a Successful First Attempt Placement
Description: The number of patients in whom the assigned device was successfully placed in the first attempt as per protocol.
Time Frame: Time taken for successful placement
Population: As per protocol,of all the patients intubated with the assigned specific device number of patients in whom the device was placed successfully in the first attempt.
Measure: Number; unit: Participants
Arm/Group | Disposable Laryngeal Tube Suction (LTS-D) | Esophageal Tracheal Combitube(ETC) | ProSeal Laryngeal Mask Airway (PLMA)
Number analyzed (Participants) | 73 | 73 | 72
Participants | 65 | 49 | 52

3. Primary Outcome: Number of Patients Who Required Multiple Attempts.
Description: The number of repeated attempts required for successfully placing the device. Each device was given a chance of 3 attempts if still unsuccessful after 3 attempts another device was placed.
Time Frame: Time taken for intubation
Population: As per protocol,the number of cases in whom the device could not be placed successfully in first attempt and required 2nd and 3rd attempts.
Measure: Number; unit: Participants
Arm/Group | Disposable Laryngeal Tube Suction (LTS-D) | Esophageal Tracheal Combitube(ETC) | ProSeal Laryngeal Mask Airway (PLMA)
Number analyzed (Participants) | 73 | 73 | 72
Participants | 8 | 24 | 20
Statistical Analysis 1: Comparison: Disposable Laryngeal Tube Suction (LTS-D) vs ProSeal Laryngeal Mask Airway (PLMA); Test type: Superiority or Other; p = 0.013, Regression, Logistic; Logistic regression Number of obs = 217, LR chi2(2)=10.89, Prob>chi2=0.0043,Log likelihood = -112.87788, Pseudo R2=0.0460; Odds Ratio (OR) = 3.125, 95% CI [1.27 to 7.67] — this is a simple odds ratio
Statistical Analysis 2: Comparison: Disposable Laryngeal Tube Suction (LTS-D) vs Esophageal Tracheal Combitube(ETC); Test type: Superiority or Other; p = 0.003, Odds ratio; Odds Ratio (OR) = 3.81, 95% CI [1.57 to 9.29]

4. Primary Outcome: Leak Pressures
Description: The maximum leak pressure attained for each device.
Time Frame: Duration of surgery
Measure: Mean (Standard Deviation); unit: cm of H2O
Arm/Group | Disposable Laryngeal Tube Suction (LTS-D) | Esophageal Tracheal Combitube(ETC) | ProSeal Laryngeal Mask Airway (PLMA)
Number analyzed (Participants) | 73 | 73 | 72
cm of H2O | 25.9 (4.6) | 23.5 (5.3) | 24.4 (5.09)
Statistical Analysis 1: Comparison: Disposable Laryngeal Tube Suction (LTS-D) vs Esophageal Tracheal Combitube(ETC); Test type: Superiority or Other; p = 0.006, t-test, 2 sided; Odds Ratio (OR) = 0.006

5. Primary Outcome: Post Operative Morbidity
Description: We followed the patients 2 and 24 hours after the surgery for sore throat, hoarseness and dysphagia.The numbers represented here are the number of patients who reported sore throat at 2 hrs and after 24 hrs as per the protocol.
Time Frame: 2 hrs and 24 hrs after surgery
Population: As per protocol,all the patients were followed up at 2 hrs and 24hrs to check for any postoperative hoarseness, sorethroat and difficulty swallowing. The numbers represent the number of patients who complained of postoperative morbidity.
Measure: Number; unit: participants
Arm/Group | Disposable Laryngeal Tube Suction (LTS-D) | Esophageal Tracheal Combitube(ETC) | ProSeal Laryngeal Mask Airway (PLMA)
Number analyzed (Participants) | 73 | 73 | 72
participants | 10 | 39 | 5
Statistical Analysis 1: Comparison: Disposable Laryngeal Tube Suction (LTS-D) vs Esophageal Tracheal Combitube(ETC); Test type: Superiority or Other; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 5.088, 95% CI [1.728 to 14.99]
Statistical Analysis 2: Comparison: Esophageal Tracheal Combitube(ETC) vs ProSeal Laryngeal Mask Airway (PLMA); Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 7.22, 95% CI [2.419 to 21.527]

6. Primary Outcome: Number of Failed Cases
Description: We calculated the number of failed cases. As per protocol, that is number of patients in whom successful intubation was not achieved with the assigned device after 3 attempts.
Time Frame: Time taken for successful intubation
Population: As per protocol, a case is decided as a failed case when the patient was not able to be intubated with the assigned device after 3 attempts.
Measure: Number; unit: Participants
Arm/Group | Disposable Laryngeal Tube Suction (LTS-D) | Esophageal Tracheal Combitube(ETC) | ProSeal Laryngeal Mask Airway (PLMA)
Number analyzed (Participants) | 73 | 73 | 72
Participants | 4 | 9 | 5

ADVERSE EVENTS:
Arm/Group | Disposable Laryngeal Tube Suction (LTS-D) | Esophageal Tracheal Combitube(ETC) | ProSeal Laryngeal Mask Airway (PLMA)
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/73 | 0/72
Other Adverse Events (participants affected / at risk) | 0/73 | 0/73 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No